CLINICAL TRIAL: NCT04115085
Title: Study of Medical Ultrasound for Rhizarthrosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Waldfriede Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUR
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Rhizarthrosis
Keywords: Degeneration; Trapeziometacarpal osteoarthritis; Basal Joint Arthritis; Arthrosis; Hand; Thumb
MeSH Terms: conditions — Osteoarthritis | interventions — Ultrasonic Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hand therapy (Experimental): 9 weeks of standard hand therapy including two 20 min slots per week.
  Interventions: Procedure: Hand therapy (18 treatments)
- Therapeutic ultrasound (Experimental): 9 weeks of standard ultra sound therapy including two 10 min slots per week.
  Interventions: Procedure: Therapeutic ultrasound (18 treatments)
- Combined hand therapy and therapeutic ultrasound (Experimental): 9 weeks of standard hand therapy plus therapeutic ultrasound including two 30 min slots per week.
  Interventions: Procedure: Combined hand therapy and therapeutic ultrasound (18 treatments)
- Sham ultrasound group (Sham Comparator): 9 weeks of sham ultrasound therapy including two 10 min slots per week.
  Interventions: Procedure: Sham ultrasound group (18 treatments)

INTERVENTIONS:
Procedure: Hand therapy (18 treatments) — 18 treatments (ea. 20 Min) within 9 weeks
  Arms: Hand therapy
Procedure: Therapeutic ultrasound (18 treatments) — 18 treatments (ea. 10 Min) within 9 weeks
  Arms: Therapeutic ultrasound
Procedure: Combined hand therapy and therapeutic ultrasound (18 treatments) — 18 treatments (ea. 30 Min) within 9 weeks
  Arms: Combined hand therapy and therapeutic ultrasound
Procedure: Sham ultrasound group (18 treatments) — Sham ultrasound group receive 18 treatments (ea. 10 Min) within 9 weeks
  Arms: Sham ultrasound group

SUMMARY:
It was never investigated which preservative non-invasive treatments are superior to treat rhizarthrosis. This randomized study compares the effect of 1. hand therapy vs. 2. therapeutic ultrasound vs. 3. hand therapy plus therapeutic ultrasound in the treatment of rhizarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40 to 90 years
* Pain intensity in the region of the thumb base in pain phases ≥ 40 mm on the VAS of 0 to 100 mm (relative to the last 24 hours)
* Complaints for at least 3 months
* X-ray Stadium Eaton I-IV at least once secured

Exclusion Criteria:

* History of surgery on the affected hand, wrist or forearm
* Planned surgery in the next 8 months
* Anticoagulation (Marcumar, Heparin)
* Haemophilia, V. Willebrandt Jürgens syndrome, thrombocytopathy and other blood anomalies
* acute pain medication (<7 days)
* Systemic medication with corticoids or immunosuppressants
* Intraarterticular injections or RSO within the last 3 months
* Pregnancy, lactation
* Insulin-dependent type I diabetes mellitus
* Significant cognitive impairment
* clinically relevant or progressive disease (e.g., liver, kidney, cardiovascular system, respiratory tract, vascular system, brain, metabolism, thyroid) that could affect the course of the study
* Malignant disease
* Simultaneous participation in an interventional study or participation in an interventional study in the last two months before study inclusion
* Clinically relevant addiction or substance abuse disorder (defined as alcohol, drug and drug abuse)
* Insufficient mental possibility of cooperation
* Therapy with oral anticoagulants (e.g., Marcumar)
* Suspected lack of compliance
* Medical, psychiatric or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or to complete the study

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | Change after 9 weeks and 3, 4 and 8 months
  Disabilities as measured by the DASH scale; No Difficulty (1), Mild Difficulty (2), Moderate Difficulty (3), Severe Difficulty (4), Unable (5)

SECONDARY OUTCOMES:
Visual analogue scale (VAS) pain | Change after 9 weeks and 3, 4 and 8 months
  From 0mm (no pain) to 100mm (maximum pain imaginable)
Short Form 36 SF-36 | Change after 9 weeks and 3, 4 and 8 months
  Scored review of health questionnaire
Functional assessment: Thumb force | Change after 9 weeks and 3, 4 and 8 months
  Key pinch force measure of the thumb as measured in Kg.
Functional assessment: Goniometry | Change after 9 weeks and 3, 4 and 8 months
  Measurement of the angle between the dorsal axis of the thumb and the index finger with a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Bock, Dr. med., Principal Investigator — Waldfriede Hospital; Martin Lautenbach, Dr. med., Study Chair — Waldfriede Hospital
Locations (1):
- Waldfriede Hospital, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bock M, Eisenschenk A, Lorenzen H, Lautenbach M. Study of Medical Ultrasound for Rhizarthrosis (SUR): study protocol for a randomized controlled single-center pilot-trial. Trials. 2020 Jun 1;21(1):450. doi: 10.1186/s13063-020-04375-2. PMID 32487163